CLINICAL TRIAL: NCT05882253
Title: Validation, Calibration, and Translation of Restriction Spectrum Imaging Signal Maps to Enhance MRI Diagnostic Capabilities in Prostate Cancer
Brief Title: Prostate Cancer IMAGing IN Early Detection (IMAGINED Trial)
Acronym: IMAGINED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mivchael Liss, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC20220897H; R01CA279667 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Detection of prostate cancer; software application
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who have agreed to undergo an MRI and subsequent prostate needle biopsy will be approached to participate in the trial. The patient will undergo the prostate MRI as standard of care. The OnQ Prostate will be acquired at the same time as the standard of care MRI at no additional cost to the subject. The MRI images will be acquired using MRI equipment manufactured by 3 different companies, depending on which facility they have their imaging performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MRI imaging using Siemens MRI (Other): Participants enrolled will undergo routine Magnetic Resonance Imaging (MRI) to obtain Restricted Spectrum Mapping (RSM). These sequences are acquired at the same time as standard multi-parametric MRI sequences. Second post-processing software then transfers the acquired RSI images from DICOM format and applies a color-coded image that is then overlayed onto the anatomic T2 image.
  Interventions: Other: Restricted Spectrum Imaging-Magnetic Resonance Imaging (RSI-MRI)
- MRI imaging using Phillips MRI (Other): Participants enrolled will undergo routine MRI to obtain RSM. These sequences are acquired at the same time as standard multi-parametric MRI sequences. Second post-processing software then transfers the acquired RSI images from DICOM format and applies a color-coded image that is then overlayed onto the anatomic T2 image.
  Interventions: Other: Restricted Spectrum Imaging-Magnetic Resonance Imaging (RSI-MRI)
- MRI imaging using General Electric (GE) MRI (Other): Participants enrolled will undergo routine MRI to obtain RSM. These sequences are acquired at the same time as standard multi-parametric MRI sequences. Second post-processing software then transfers the acquired RSI images from DICOM format and applies a color-coded image that is then overlayed onto the anatomic T2 image.
  Interventions: Other: Restricted Spectrum Imaging-Magnetic Resonance Imaging (RSI-MRI)

INTERVENTIONS:
Other: Restricted Spectrum Imaging-Magnetic Resonance Imaging (RSI-MRI) — An advanced imaging software that supports improved prostate cancer detection and diagnosis
  Other Names: On-Q Prostate

SUMMARY:
The researchers hope to learn if specific types of MRI software and techniques can help improve early prostate cancer detection at time of a MRI-guided prostate biopsy.

DETAILED DESCRIPTION:
A phase 2 prospective, interventional, non-randomized clinical trial design to investigate whether Restricted Spectrum Maps (RSM) attained from RSI-MRI (On-Q Prostate) improves PI-RADS accuracy compared to PI-RADS alone for the detection of clinically significant prostate cancer. Patients who have agreed to undergo an MRI and subsequent prostate needle biopsy will be approached to participate in the trial.

The aims of the study are as follows:

Goal 1. Validate RSI-MRI imaging biomarker performance using a prospective clinical trial.

Goal 2. Calibrate the RSM values across different MRI scanner manufacturers. Goal 3. Translate RSI using a net clinical benefit model.

ELIGIBILITY:
Inclusion Criteria:

* Selected to undergo an MRI-fusion prostate needle biopsy of the prostate.
* Able to provide informed consent

Exclusion Criteria:

* prior diagnosis of prostate cancer (Grade Group >1)
* metastatic prostate cancer
* prior prostate cancer treatment
* contraindication to prostate biopsy (e.g., on anticoagulation that cannot be safely discontinued)
* inability to undergo MRI (e.g., too large to be accommodated in a scanner or with an implant incompatible with MRI).
* Bilateral hip replacement
* Unable to provide informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
RSM mapping value | Baseline to approximately 9 months
  Radiologists will report a standard Prostate Imaging, Reporting, and Data System (PI-RADS) and document the RSM values associated with each lesion. Change in value will be reported from baseline to routine biopsy follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Liss, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers